CLINICAL TRIAL: NCT01959815
Title: Novel Screening Strategies for Scleroderma PAH (Pulmonary Arterial Hypertension)
Brief Title: Novel Screening Strategies for Scleroderma PAH
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Scott Visovatti, MD, Assistant Professor, University of Michigan
Other Study IDs: HUM00074818
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Arterial Hypertension; Scleroderma
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Blood samples will be drawn at rest and during exercise.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Scleroderma and diagnosed PAH
- "Low risk" scleroderma
- Healthy volunteers
- "High risk" scleroderma

SUMMARY:
Patients with scleroderma can develop heart failure due to high blood pressure in the lungs (a condition called pulmonary arterial hypertension). It is important to find pulmonary arterial hypertension early, so that it can be treated before heart failure develops. However, the tests that we now use to find the earliest form of this disease in scleroderma patients are not good enough. This study will examine whether tests performed during exercise can improve our ability to find early pulmonary arterial hypertension. The study will also try to identify genes that are responsible for the development of pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 30 years or older;
* diagnosis of limited or diffuse scleroderma (American College of Rheumatology criteria)
* for the "high risk" group, one of the following features:

  * resting transthoracic echocardiogram showing elevated right-sided pressures within previous 3 months [tricuspid regurgitation (TR) jet >2.8 m/s or evidence of right ventricular dysfunction]
  * pulmonary function testing (PFT) showing abnormal diffusing capacity of carbon monoxide (DLCO) not due to significant interstitial lung disease (DLCO<60% predicted or FVC: DLCO ratio >1.4)

Exclusion Criteria:

* Pregnancy
* prior diagnosis of pulmonary hypertension
* treatment with endothelin receptor antagonists, phosphodiesterase-5 inhibitors, or prostacyclin analogues
* previous diagnosis of obstructive lung disease or pulmonary thromboembolic disease
* current smoker
* significant valvular disease
* resting echocardiogram showing left ventricular ejection fraction<50% within previous 3 months
* resting echocardiogram showing significant (greater than Grade I) diastolic dysfunction
* pulmonary emboli (past or present).

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers will be recruited from scleroderma clinics, pulmonary hypertension clinics, and (for healthy volunteers) the Ann Arbor area.
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2013-09-26 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-11-06 (Actual)

PRIMARY OUTCOMES:
Development of pulmonary arterial hypertension | Two years after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Scott H Visovatti, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States